CLINICAL TRIAL: NCT06884670
Title: Assessment of Efficacy and Safety of PD-1 Monoclonal Antibody Combined With IL-2 and CapeOX in Neoadjuvant Therapy for Locally Advanced Rectal Cancer Prior to Surgery: A Prospective, Multi-center, Randomized Controlled Study (PICM)
Brief Title: Assessment of Efficacy and Safety of PD-1 Monoclonal Antibody Combined With IL-2 and CapeOX in Neoadjuvant Therapy for Locally Advanced Rectal Cancer Prior to Surgery: A Prospective, Multi-center, Randomized Controlled Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICM
Record Dates: First submitted 2024-07-11; First posted 2025-03-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer
Keywords: Tislelizumab; Interleukin-2; MSS/pMMR rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Interleukin-2; Radiotherapy; tislelizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Neoadjuvant Group (Active Comparator): Radiotherapy 1.8Gy per time*28 And Capecitabine: 825mg/m2 bid po, a total of 28 days CapeOX 2 cycles (Capecitabine: 825mg/m2 bid po, d1-d14；Oxaliplatin 200 mg/m² ivd, d1
  Interventions: Radiation: Radiotherapy; Drug: Oxaliplatin; Drug: Capecitabine
- PD-1+IL-2+CapeOX group (Experimental): Tislelizumab 200mg ivd D1+Interleukin 2 100IU HD, d1-d14+ CapeOX (total 6 cycles)
  Interventions: Drug: Interleukin-2; Drug: Tislelizumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Interleukin-2 — Tislelizumab 200mg ivd D1+Interleukin 2 100IU HD, d1-d14+ CapeOX (Capecitabine: 825mg/m2 bid po, d1-d14；Oxaliplatin 200 mg/m² ivd, d1)
  Arms: PD-1+IL-2+CapeOX group
Radiation: Radiotherapy — Radiotherapy 1.8Gy per time*28
  Arms: Conventional Neoadjuvant Group
Drug: Tislelizumab — Tislelizumab 200mg ivd D1
  Arms: PD-1+IL-2+CapeOX group
Drug: Oxaliplatin — Oxaliplatin 200 mg/m² ivd, d1
Drug: Capecitabine — Capecitabine: 825mg/m2 bid po, d1-d14

SUMMARY:
The objective is to evaluate whether the neoadjuvant combination of tislelizumab (a PD-1 inhibitor) with interleukin-2 (IL-2) chemotherapy can significantly increase the Objective Response Rate (ORR) and the Pathological Complete Response rate (pCR) in patients with locally advanced rectal cancer who have Microsatellite Stable/Proficient Mismatch Repair (MSS/pMMR) status.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) stands as a prominent global health concern, ranking among the most prevalent malignancies worldwide. Its incidence exhibits striking geographical variations, with higher rates observed in developed countries. Age is a significant risk factor, predominantly affecting individuals aged 50 and above, although a concerning trend of increasing incidence in younger adults has been noted in recent years. There exists a gender disparity, with slightly higher prevalence in males. Notably, lifestyle factors, including dietary choices, sedentary habits, smoking, and obesity, play crucial roles in its etiology. These epidemiological patterns underscore the urgency for implementing effective prevention strategies and advancing early detection methods to mitigate the disease's impact.

In recent years, substantial advancements have reshaped the landscape of CRC treatment, offering new hope and improved outcomes for affected individuals. Surgical intervention remains the cornerstone of curative therapy, guided by tumor stage, location, and patient's overall health status. Adjuvant therapies, including chemotherapy and radiotherapy, have been pivotal in reducing recurrence rates and enhancing overall survival. Targeted treatments, such as anti-EGFR and anti-VEGF drugs, have ushered in an era of precision medicine, selectively targeting critical molecular pathways. Meanwhile, immunotherapy, particularly immune checkpoint inhibitors, has emerged as a promising frontier, offering personalized treatment options for CRC patients.

In CRC, the PD-1 inhibition pathway plays a central role in regulating immune cell exhaustion; however, the response to PD-1 monotherapy is limited in a majority of colorectal cancer patients, suggesting that combining PD-1 blockade with other immunostimulatory agents holds promise. Currently, several combination therapies have shown progress in animal models and are being explored in clinical studies. Among these, interleukin-2 (IL-2) emerges as a candidate drug, synergizing with PD-1 blockade to potentiate antitumor effects. This study aims to investigate the combination of IL-2 with PD-1 inhibitors, seeking to overcome the limitations of single-agent immunotherapy through multifaceted immunomodulation. By modulating the immune microenvironment to enhance immune cell infiltration and break down the physical and immunosuppressive barriers of the tumor, this approach seeks to augment the efficacy of immunotherapy, particularly for immunologically cold CRC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged between 18 and 75 years;
2. An Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
3. Histologically confirmed rectal adenocarcinoma;
4. Clinical stage T3-T4 or any T with node-positive (N+) disease: locally advanced;
5. Microsatellite stable (MSS) status;
6. Adequate hematological, hepatic, and renal functions.

Exclusion Criteria:

1. Patients with metastatic disease (Stage IV); recurrent colorectal cancer with active bleeding, perforation, or complex conditions requiring urgent surgery; or concurrent non-colorectal cancer malignancies.
2. Patients who have previously received systemic anticancer therapy for colorectal cancer; or have been treated with PD-1, PD-L1, or CTLA-4 antibodies.
3. Patients with any active autoimmune disease; known or tested positive for Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS); or a history requiring steroid or immunosuppressive drug treatment.
4. Patients with interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases (such as diabetes, hypertension, pulmonary fibrosis, and acute pneumonia).
5. Patients who experienced any Grade 2 or higher toxicities due to prior treatments (as classified by the Common Terminology Criteria for Adverse Events [CTCAE] version 5), which have not resolved (excluding anemia, alopecia, and skin pigmentation changes); known or suspected history of hypersensitivity to any of the drugs used in the trial.
6. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 1 years
Pathological Complete Response rate (pCR) | 1 year
Clinical complete response (cCR) | 1 years

SECONDARY OUTCOMES:
Safety and Tolerability | 1 month

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Nanjing BenQ Hospital, Nanjing, Jiangsu
  - Jiangsu province hospital, Nanjing, Jiangsu
  - Xuzhou Central hospital, Xuzhou, Jiangsu
  - The Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided